CLINICAL TRIAL: NCT04467593
Title: A Mono-centric, First In-human (FIH), Safety and Preliminary Efficacy Study of (Neo)Adjuvant, Model-based, Whole-body Hyperthermia (WBHT) Treatment in Advanced Solid Cancer Patients or Stage IV (TxNxM1) Metastatic Pancreatic Adenocarcinoma Patients
Brief Title: Safety Study of Whole Body Hyperthermia for Advanced Cancer
Acronym: MATTERS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElmediX (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MATTERS 1
Record Dates: First submitted 2020-06-24; First posted 2020-07-13 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Advanced Cancer; Pancreatic Cancer Metastatic
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort A1 (Experimental): Three patients with advanced solid cancer will be subjected to repetitive hyperthermia starting with 2 hours (day 1), 4 hours (day 8) and 6 hours (day 15)
  Interventions: Device: Whole body hyperthermia
- Cohort A2 (Experimental): One patient with advanced solid cancer will receive 3 hyperthermia treatments of 4 hours per treatment. The next patient with advanced solid cancer will receive 3 hyperthermia treatments of 6 hours per treatment.
  Interventions: Device: Whole body hyperthermia
- Cohort B (Experimental): Three pancreatic cancer patients will be subjected to three hyperthermia treatments (2 hours duration per treatment) alone (1st treatment) or in combination with (2nd and 3rd treatment) Standard of Care (SOC) chemotherapy according to the NCCN guidelines.
  Interventions: Device: Whole body hyperthermia; Drug: Standard of Care (SOC) chemotherapy according to the NCCN guidelines.
- Cohort C (Experimental): Three pancreatic cancer patients will be subjected to three hyperthermia treatments (4 hours duration per treatment) alone (1st treatment) or in combination with (2nd and 3rd treatment) Standard of Care (SOC) chemotherapy according to the NCCN guidelines.
  Interventions: Device: Whole body hyperthermia; Drug: Standard of Care (SOC) chemotherapy according to the NCCN guidelines.
- Cohort D (Experimental): Three pancreatic cancer patients will be subjected to three hyperthermia treatments (6 hours duration per treatment) alone (1st treatment) or in combination with (2nd and 3rd treatment) Standard of Care (SOC) chemotherapy according to the NCCN guidelines.
  Interventions: Device: Whole body hyperthermia; Drug: Standard of Care (SOC) chemotherapy according to the NCCN guidelines.

INTERVENTIONS:
Device: Whole body hyperthermia — Whole body hyperthermia to treat stage IV cancer patients
Drug: Standard of Care (SOC) chemotherapy according to the NCCN guidelines. — Whole body hyperthermia to treat stage IV pancreatic cancer patients combined with standard of care chemotherapy
  Arms: Cohort B; Cohort C; Cohort D

SUMMARY:
Millions of patients die of cancer every year. There are several methods to treat cancer, including surgery, chemotherapy, radiotherapy and immunotherapy. Recently, hyperthermia therapy started playing a role in cancer therapy. It has shown effect in animal experiments and clinical practice. The sponsor has developed a novel device to use hyperthermia for advanced cancer. This study is to prove the safety in human patients of this device & therapy and get the first data on efficacy.

ELIGIBILITY:
Inclusion criteria:

1. Patients between 18- and 75-years of age at time of signing the informed consent
2. Patients with advanced solid cancer (for cohort A1, A2 only) or metastatic pancreatic adenocarcinoma confirmed by histology (for cohort B/C/D only)
3. Patients previously treated or under treatment with standard of care treatment (cohort B/C/D only) or patients without treatment options
4. WHO performance status ≤ 1(see appendix V)
5. Maximum waist circumference ≤ 150 cm
6. Weight ≤ 100 kg
7. Height ≤ 1,90 m
8. Adequate liver structure (confirmed by CT scan) allowing the placement of the liver sensor
9. No (prostate) pathology that would interfere with the placement of the bladder catheter
10. Adequate bone marrow function defined as

    1. white blood cell count ≥ 2000/µl
    2. neutrophils ≥ 1500 cells/μL
    3. platelets ≥ 100 x 109/L
    4. hemoglobin ≥ 10 g/dl documented within 1 week prior to first treatment
11. Adequate coagulation defined as

    1. PT (%) ≥ 70%
    2. aPTT ≤ ULN
    3. Von Willebrand Factor Antigen ≥ LLN
    4. Von Willebrand Factor Activity ≥ LLN
    5. PFA COL/EPI CT ≤ 1.15 ULN
    6. PFA COL/ADP CT ≤ 1.15 ULN
12. Adequate liver function defined as

    1. Transaminases (AST, ALT) ≤ 2.5 x ULN or ≤ 5.0 in presence of liver metastasis
    2. bilirubin ≤ 2 x ULN documented
13. Adequate renal function defined as

    1. serum creatinine ≤ 1.6 mg/dL (male); ≤ 1.3 mg/dL (female);
    2. albumin ≥ 30g/L
    3. calculated eGFR ≥ 60 mL/min (CKD-EPI equation) documented within 1 week prior to randomization
14. No blood donation 3 months prior to the WBHT treatment
15. No participation in other clinical trial 4 weeks prior to the WBHT treatment
16. No biological therapy 4 weeks prior to the WBHT treatment or during WBHT treatment
17. No surgery 4 weeks prior to the WBHT treatment
18. No radiotherapy 3 weeks prior to the WBHT treatment or during WBHT treatment
19. No chemotherapy 1 week prior to the WBHT treatment (for cohort A/B/C/D) or during WBHT treatment (for Cohort A1/A2)
20. No anti-platelet aggregation medication intake from 5 days prior to the first WBHT treatment until 5 days after the last treatment
21. No anticoagulant medication intake between screening and last follow-up visit. However, if deemed necessary by the investigator, the patient may receive prophylactic Low Molecular Weight Heparin on the day prior to the first WBHT treatment until 10 days after the last WBHT treatment
22. No transdermal patches during participation in the study
23. No piercings (internally or externally)during WBHT treatment
24. Life expectancy of at least 18 weeks
25. Effective contraception for both male and female patients if applicable. Women of childbearing potential must have negative blood pregnancy test at screening visit.
26. Written informed consent must be given according to good clinical practice and national/local regulations.

Exclusion criteria:

1. Pregnant or breastfeeding women (based on HCG levels)
2. Presence of brain metastasis (known or suspected)
3. Other malignant diseases in the medical history during the last 5 years (exceptions: carcinoma in situ of the cervix or adequately treated basal cell carcinoma of the skin)
4. Serious medical risk factors involving any of the major organ systems, including high cardiovascular risk, coronary stenting or myocardial infarction in the last year
5. Clinically significant pulmonary disease which might interfere with mechanical ventilation
6. History of autonomic dysfunction (due to the influence on skin blood flow)
7. History of malignant hyperthermia or a positive diagnostic test (Caffeine-Halothane Contracture test) in case of family history of malignant hyperthermia.
8. History of untreated endocrine pathology (e.g. diabetes type II, hyper- or hypothyroidism).
9. Primary diabetes type I (due to vascular complications)
10. Known allergies to drugs that will be used during the trial (e.g. anesthetic, analgesic, (chemotherapy used in cohort B/C/D))
11. Active infections not controlled by medication
12. Severe, non-healing wounds, ulcers or bone fractures
13. Organ allografts requiring immunosuppressive therapy
14. (History of) clinically significant (investigator decision) psychiatric disorder and/or psychosocial disorder that may interfere with adequate compliance to the protocol or signature of the informed consent
15. Other clinically significant disease which could impair the patient's ability to participate in the study according to the investigator's opinion
16. Participation in another clinical trial during this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse device events (ADEs) in relation to the medical device | 4 weeks after last treatment
Incidence of related clinically significant abnormalities on electrocardiogram (ECG), vital signs, physical examination and laboratory parameters | 4 weeks after last treatment
Incidence of adverse events (AEs) related to WBHT treatment alone or in combination with SOC chemotherapy according to the NCCN guidelines. nab-paclitaxel or gemcitabine alone | 4 weeks after last treatment

SECONDARY OUTCOMES:
evolution of CA19-9 (U/ml) | 4 weeks after last treatment
  The evolution of this clinically significant biological parameter will be measured compared to baseline
evolution of CEA (ng/ml) | 4 weeks after last treatment
  The evolution of this clinically significant biological parameter will be measured compared to baseline
based on the three primary outcome measures, guidance will be drafted for phase II treatment duration in combination with chemotherapy dosing. | 4 weeks after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Marc Peeters, MD PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Edegem, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No